CLINICAL TRIAL: NCT05931718
Title: Evaluation of the Diagnostic/Therapeutic Course of Patients With Autoimmune Cytopenias (Autoimmune Hemolytic Anemia AIHA, Immune Thrombocytopenia ITP, Chronic Idiopathic/Autoimmune Neutropenia CIN/AIN) and Identification of Predictive and Prognostic Markers.
Brief Title: Prospective Evaluation of Diagnosis and Treatment of Patients With Autoimmune Cytopenias Including Autoimmune Hemolytic Anemia, Immune Thrombocytopenia, and Chronic Idiopathic/Autoimmune Neutropenia
Acronym: AIHA ITP CIN
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: CYTOPAN
Record Dates: First submitted 2023-05-29; First posted 2023-07-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Autoimmune Hemolytic Anemia; Immune Thrombocytopenia; Chronic Idiopathic Neutropenia; Autoimmune Neutropenia; Myelodysplastic Syndromes; Cold Agglutinin Disease
Keywords: autoimmune hemolytic anemia; immune thrombocytopenia; chronic idiopathic neutropenia; autoimmune neutropenia; cold agglutinin disease; myelodysplastic syndromes; rituximab; thrombopoietin receptor agonists; erythropoietin; steroids; splenectomy; red cell metabolism; cytokines; luspatercept; microbiome; single cell analysis; next generation sequencing
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Purpura, Thrombocytopenic, Idiopathic; Myelodysplastic Syndromes | interventions — Fecal Microbiota Transplantation; Erythropoietin; luspatercept; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood for cytokines and next generation sequencing, bone marrow sample for single cell analysis, fecal sample for microbiome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Autoimmune hemolytic anemia: AIHA patients will be enrolled at diagnosis and stratified according to AIHA type (i.e. warm, cold, mixed, and atypical forms), sampled for peripheral blood for cytokine and NGS studies, and for feces for microbiome studies. If clinically indicated, bone marrow evaluation will be performed and a sample for single cell analysis will be collected. Patients will be followed up to collect treatments, responses, relapses, and complications (particularly thromboses and infections).
  Interventions: Biological: cytokine essays; Biological: NGS; Biological: Fecal microbiome; Drug: Erythropoietin
- Immune thrombocytopenia: ITP patients will be enrolled at diagnosis and sampled for peripheral blood for cytokine and NGS studies, and for feces for microbiome studies. If clinically indicated, bone marrow evaluation will be performed and a sample for single cell analysis will be collected.Patients will be followed up to collect treatments, responses, relapses, and complications (particularly thromboses and infections).
  Interventions: Biological: cytokine essays; Biological: NGS; Biological: Fecal microbiome; Drug: Thrombopoietin Receptor Agonist
- Chronic idiopathic neutropenia/Autoimmune neutropenia: CIN/AIN patients will be enrolled at diagnosis and sampled for peripheral blood for cytokine and NGS studies, and for feces for microbiome studies. If clinically indicated, bone marrow evaluation will be performed and a sample for single cell analysis will be collected.Patients will be followed up to collect treatments, responses, relapses, and complications (particularly infections).
  Interventions: Biological: cytokine essays; Biological: NGS; Biological: Fecal microbiome; Drug: G-CSF
- Myelodysplastic syndromes: MDS patients will be enrolled at diagnosis and sampled for peripheral blood for cytokine and NGS studies, and to evaluate red cell metabolism. If clinically indicated, bone marrow evaluation will be performed and a sample for single cell analysis will be collected. Patients will be followed up to collect treatments, responses, relapses, and outcome.
  Interventions: Biological: cytokine essays; Biological: NGS; Biological: Fecal microbiome; Drug: Luspatercept

INTERVENTIONS:
Biological: cytokine essays — evaluation of immunomodulatory cytokines by ELISA kits on peripheral blood samples
Biological: NGS — evaluation of somatic mutations commonly associated with myeloid neoplasm and immunodeficiencies by next generation sequencing on peripheral blood samples
Biological: Fecal microbiome — evaluation of fecal microbiome on fecal samples
Drug: Erythropoietin — evaluation of recombinant erythropoietin use, safety and efficacy in patients with autoimmune hemolytic anemia according to clinical practice
  Groups: Autoimmune hemolytic anemia
Drug: Luspatercept — evaluation of cytokine levels, molecular profile and bone marrow microenvironment by single cell analysis in patients treated with luspatercept according to clinical practice
  Groups: Myelodysplastic syndromes
Drug: Thrombopoietin Receptor Agonist — evaluation of TPO-RA use, safety and efficacy in patients with ITP according to clinical practice
  Groups: Immune thrombocytopenia
Drug: G-CSF — evaluation of G-CSF use, safety and efficacy in patients with CIN/AIN according to clinical practice
  Groups: Chronic idiopathic neutropenia/Autoimmune neutropenia

SUMMARY:
The goal of this observational study is to characterize the diagnostic and therapeutic management of autoimmune cytopenias including autoimmune hemolytic anemia, immune thrombocytopenia, and chronic idiopathic/autoimmune neutropenia.

The main aims to answer are:

* evaluation of traditional and novel diagnostic tools including immunohematology, cytokine essays, bone marrow studies, molecular findings, and fecal microbiome.
* evaluation of type and sequence of the therapies administered, the response rates, and the adverse events.
* evaluation of clinical and laboratory (immunologic, molecular, and morphologic) predictors of outcome.
* evolution of autoimmune cytopenias into myelodysplastic syndromes.
* a subgroup of patients with myelodysplastic syndromes will be included to evaluate the presence of immunologic events, autoimmune activation, and red cell metabolism.

Participants will receive a clinical/laboratory diagnostic workup as per current clinical practice. Furthermore They will be sampled at baseline (peripheral blood and feces for microbiome) and followed up for at least 3 years to evaluate their clinical course, therapeutic management and outcome.

DETAILED DESCRIPTION:
This observational study will characterize the diagnostic and therapeutic management of autoimmune cytopenias including autoimmune hemolytic anemia, immune thrombocytopenia, and chronic idiopathic/autoimmune neutropenia to evaluate predictors of outcome. Additionally, a subgroup of patients with myelodysplastic syndromes (diagnosed according to current WHO 5th edition 2022) will be included to evaluate the presence of autoimmune activation, and red cell metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autoimmune cytopenias (AIHA/ITP/CIN/AIN)
* age >/= 18 years
* ability to sign informed consent
* availability to undergo 3 year follow up
* for the subgroup of patients with myelodysplastic syndrome: bone marrow evaluation showing >/= 10% dysplastic features of at least one lineage along with MDS defining cytopenia and/or MDS defining cytogenetics.

Exclusion Criteria:

* any condition impeding the acquisition of the informed consent
* immune cytopenia diagnosis preceding >/= 6 months the enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anemia (Hb <12 g/dL), thrombocytopenia (PLT<100.000/mmc) and/or neutropenia (neutrophils<1000/mmc) attending the inpatient or outpatient facility of Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy.
  Cytopenia diagnosis will be based on current guidelines for AIHA (evidence of hemolysis and positive direct Coombs test or negative once excluded other causes), for ITP (exclusion of other thrombocytopenia causes) and for CIN/AIN (exclusion of other neutropenia causes). Patients will be classified according to the degree of the cytopenia and, for AIHA, according to thermal characteristics (warm, cold, mixed, atypical).
  For the substudy of patients with MDS patients will be stratified according to WHO 2022 classification of myeloid neoplasms.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
sensitivity of autoantibody testing in autoimmune cytopenias | 2021-2026
  to define the sensitivity of autoantibody testing in autoimmune cytopenias
specificity of autoantibody testing in autoimmune cytopenias | 2021-2026
  to define the specificity of autoantibody testing in autoimmune cytopenias
sensitivity of bone marrow trephine in autoimmune cytopenias | 2021-2026
  to define the sensitivity of bone marrow trephine in autoimmune cytopenias

SECONDARY OUTCOMES:
overall response rate | 2021-2026
  to define response rates to treatment of autoimmune cytopenias and myelodysplastic syndromes
Evaluation of somatic mutations | 2021-2026
  to define somatic mutations in autoimmune cytopenias and myelodysplastic syndromes by NGS
Evaluation of pyruvate kinase activity | 2021-2026
  to define pyruvate kinase activity in myelodysplastic syndromes
Evaluation of microbiome | 2021-2026
  to define microbiome composition in autoimmune cytopenias and myelodysplastic syndromes
Single cell RNA expression | 2021-2026
  to define bone marrow composition by single cell analysis in autoimmune cytopenias and myelodysplastic syndromes
Evaluation of cytokine levels | 2021-2026
  to define cytokine levels in autoimmune cytopenias and myelodysplastic syndromes by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fattizzo B, Pedone GL, Brambilla C, Pettine L, Zaninoni A, Passamonti F, Barcellini W. Recombinant erythropoietin in autoimmune hemolytic anemia with inadequate bone marrow response: a prospective analysis. Blood Adv. 2024 Mar 12;8(5):1322-1327. doi: 10.1182/bloodadvances.2023011798. PMID 38029356
- [Derived] Versino F, Revelli N, Villa S, Pettine L, Zaninoni A, Prati D, Passamonti F, Barcellini W, Fattizzo B. Transfusions in autoimmune hemolytic anemias: Frequency and clinical significance of alloimmunization. J Intern Med. 2024 Mar;295(3):369-374. doi: 10.1111/joim.13753. Epub 2023 Nov 27. PMID 38013593